CLINICAL TRIAL: NCT03626649
Title: A Prospective Single Arm Clinical Evaluation for the Characterization of the Safety Profile of the DiamondTemp™ System for Fast Treatment of Patients With Atrial Fibrillation
Brief Title: Evaluation for the Characterization of the Safety Profile of the DiamondTemp™ System for Fast Treatment of Patients With Atrial Fibrillation
Acronym: FASTR-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP00983
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: The DIAMOND FASTR-AF study is a prospective, single-arm trial being performed at multiple centers in Europe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DiamondTemp Cardiac Ablation System (Experimental): Cardiac ablation procedure
  Interventions: Device: DiamondTemp Cardiac Ablation System

INTERVENTIONS:
Device: DiamondTemp Cardiac Ablation System — The DiamondTemp Ablation System is the test device in this investigational study. The DiamondTemp Ablation System consists of:
  * DiamondTemp Ablation Catheter
    o Unidirectional and Bidirectional models
  * DiamondTemp Catheter-to RFG Cable
  * DiamondTemp GenConnect Cable
  * DiamondTemp FASTR Generator with Footswitch
  * DiamondTemp Irrigation Pump
  * DiamondTemp Irrigation Tubing Set
  Other Names: Cardiac ablation

SUMMARY:
The objective of this study is to characterize the performance of the DiamondTemp Ablation System for its intended use.

DETAILED DESCRIPTION:
* The DiamondTemp Ablation System is indicated for use in patients requiring cardiac electrophysiological mapping (stimulation and recording) and, when used in conjunction with a radiofrequency generator and irrigation pump, for cardiac ablation with monitoring of tissue temperature during ablation.
* In this study, the DiamondTemp Ablation System will be evaluated for the treatment of patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for intra-cardiac mapping and ablation for arrhythmias
* History of recurrent symptomatic PAF with ≥2 episodes reported within the 365 days
* (12) months prior to enrollment
* At least 1 episode of AF documented by Holter monitor, rhythm strip, trans-telephonic monitor (TTM), or 12-lead ECG prior to enrollment
* Refractory to at least one Class I-IV anti-arrhythmic drug (AAD)
* Eighteen (18) years of age or above

Exclusion Criteria:

* Previous left atrial ablation procedure
* Intracardiac thrombus, tumor or other abnormality that precludes catheter introduction and placement
* Known severe cerebrovascular disease or history of cerebrovascular event (< 1 month)
* Subjects with severely impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR)3 with a GFR ≤ 29. Active gastrointestinal bleeding
* Active infection or fever (>100.5 F/38 ◦C)
* Sepsis
* Cardiac surgery within the past two months.
* Short life expectancy (<1 yr.) due to other illnesses, such as cancer or pulmonary, hepatic, or renal disease Significant anemia (hemoglobin < 8.0 mg/dL)
* Severe uncontrolled systemic hypertension (systolic pressure > 240 mm Hg within the last 30 days)
* Documented anaphylaxis during previous exposure to angiographic contrast media
* Uncontrolled congestive heart failure (NYHA1 Class III or IV)
* Unstable angina or acute myocardial infarction within the past three months
* Bleeding, clotting disorders, or known thrombosis
* Severe Peripheral vascular disease
* Uncontrolled diabetes
* Heart valve replacement
* Mitral clip (E-valve)
* Women who are of childbearing potential who are currently pregnant or not willing to use contraception for the duration of the study
* Active participation in another investigational protocol currently or the last 30 days
* Unable or unwilling to take anti-coagulants
* Unwilling or unable to comply with any protocol or follow up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Freedom from a composite of serious adverse events (SAE) | 30 days
  Freedom from a composite of serious adverse events (SAE)
Freedom from documented symptomatic atrial fibrillation (AF), atrial flutter(AFL) and atrial tachycardia (AT) episodes | 12 months
  Freedom from documented symptomatic atrial fibrillation (AF), atrial flutter(AFL) and atrial tachycardia (AT) episodes

SECONDARY OUTCOMES:
Freedom from a composite SAE | 7 days
  Freedom from a composite SAE
Freedom from documented symptomatic and asymptomatic AF, AT and AFL episodes | 12 months
  Freedom from documented symptomatic and asymptomatic AF, AT and AFL episodes
Rate of single procedure success | 12 months
  Rate of single procedure success

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Na Homolce
Locations (4):
- Na Homolce, Prague, Czechia
- France (3):
  - Clnique du Tonkin, Lyon
  - CHRU de Nancy, Nancy
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neuzil P, Poty H, de Chillou C, Petru J, Getman MK, Liu S, Funasako M, Durand-Dubief A, Combes S, Albenque JP. Radiofrequency ablation using the second-generation temperature-controlled diamond tip system in paroxysmal and persistent atrial fibrillation: results from FASTR-AF. J Interv Card Electrophysiol. 2023 Mar;66(2):343-351. doi: 10.1007/s10840-022-01234-9. Epub 2022 May 18. PMID 35581464